CLINICAL TRIAL: NCT06896383
Title: Role of USP35 in the Detection of Ferroptosis in Juvenile Autoimmune Hepatitis: an Immunohistochemical Study
Brief Title: Role of USP35 in the Detection of Ferroptosis in Juvenile Autoimmune Hepatitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Rashwan Mohamed, Assistant lecturer, Assiut University
Other Study IDs: USP35 in autoimmune hepatitis
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cases with juvenile autoimmune hepatitis: patients who are diagnosed physically, clinically, and histologically with juvenile autoimmune hepatitis
- control group: children with near-normal liver biopsy

SUMMARY:
1. To evaluate the immunohistochemical expression of USP35 in cases of juvenile autoimmune hepatitis and control cases.
2. To correlate this with the level of necro-inflammation and extent of fibrosis using Massion's trichrome stain in cases of juvenile autoimmune hepatitis.

DETAILED DESCRIPTION:
Autoimmune hepatitis (AIH) is a rare and chronic inflammatory disease of the liver of unknown etiology characterized by loss of immune tolerance against liver antigens leading to progressive destruction of hepatic parenchyma and if untreated leads to end-stage liver disease.

It affects all ages with a peak incidence in pediatric age, where it is referred to as Juvenile Autoimmune Hepatitis (JAIH).JAIH is a long-term condition that varies in intensity over time. It occurs more frequently in females and is marked by increased levels of serum gamma globulins, the presence of autoantibodies in the bloodstream, and interface hepatitis observed in liver histology. JAIH can occur at any age from infancy to adolescence with an incidence reported of 0.4 and a prevalence of 3.0 per 100,000 children, respectively. Diagnosing the condition can be difficult and relies on a mix of clinical, biochemical, immunological, and histological indicators, as well as ruling out any other known causes that could present similar characteristics to JAIH. Certain circulating autoantibodies are crucial indicators of the disease. AIH type 1 is characterized by anti-smooth Muscle Antibodies (SMA) and/or anti-nuclear Antibodies (ANA), AIH type 2 is defined by the detection of anti-Liver-Kidney Microsomal antibody type 1 (LKM1) and/or of anti-Liver-Cytosol antibody type 1 (LC1). Approximately 20% of children exhibiting clinical, biochemical, and histological characteristics of autoimmune hepatitis do not have either typical or atypical autoantibodies, including anti-soluble liver antigen (anti-SLA) or atypical perinuclear anti-neutrophil cytoplasmic antibody (pANCA). These individuals form a diverse category of inflammatory liver conditions referred to as "seronegative autoimmune hepatitis." A liver biopsy is frequently required to make a diagnosis in atypical situations. Histological examination helps assess the level of necro-inflammation and the extent of fibrosis. The majority of biopsies taken from children with JAIH display moderate to severe interface hepatitis and lobular inflammation. Interface hepatitis is characterized by a pronounced infiltration of mononuclear cells in the portal and periportal areas, including CD4 and CD8 T cells, macrophages, plasma cells, and, on occasion, eosinophils. Emperipolesis, which involves the infiltration of CD8 T-lymphocytes into hepatocytes, is regarded as a distinctive characteristic of autoimmune hepatitis. Its occurrence is linked to more severe necroinflammatory traits and increased levels of fibrosis.

An overview of ferroptosis:

In 2012, Dixon et al. formally named a new type of cell death as ferroptosis, according to its characteristics when studying the mechanism by which erastin killed cancer cells with RAS mutations. Ferroptosis is a new mode of cell death. Morphologically, ferroptosis presents mainly in cells as reduced mitochondrial volume, increased bilayer membrane density and reduction or disappearance of mitochondrial cristae but the cell membrane is still intact, the nucleus is normal in size, and there is no condensation of chromatin; biochemically, there is intracellular glutathione (GSH) depletion and decreased activity of glutathione peroxidase 4 (GPX4), lipid peroxides cannot be metabolized by the GPX4-catalyzed reduction reaction, and Fe2+ oxidizes lipids in a Fenton-like manner, resulting in a large amount of ROS, which induces ferroptosis and genetically, ferroptosis is a biological process regulated by multiple genes. Ferroptosis mainly includes genetic changes in iron homeostasis and lipid peroxidation metabolism, but the specific regulatory mechanism is still in a need to be further studied.As research continues, ferroptosis has been shown to be involved in the development and progression of autoimmune and inflammatory diseases.

Mechanism of ferroptosis:

Iron metabolism and ferroptosis Iron plays a necessary role in mammalian physiological processes. However, excess iron is also fatal as it catalyzes the formation of reactive oxygen species (ROS). Thus, cellular and systemic iron metabolism is intricately and tightly controlled to prevent oxidative damage caused by imbalanced iron homeostasis. Intracellular iron metabolism is a complex physiological process, and cellular homeostasis depends on normal iron metabolism. In general, the balance of intracellular iron metabolism relies on the uptake, export, and utilization of iron ions.

Iron metabolism regulates cellular sensitivity to ferroptosis by regulating the labile iron pool (LIP) . Fe3+ in the circulation maintains homeostasis of iron metabolism through tight binding and release with transferrin (TF). Fe3+ is transported by TF and enters into cells after being recognized by transferrin receptor 1 (TFR1) at cell membranes. Next, Fe3+ is reduced to Fe2+ by reductase six-transmembrane epithelial antigen of prostate 3 (STEAP3). Subsequently, divalent metal transporter 1 (DMT1) released Fe2+ into the LIP. Intracellular LIP is mainly in the form of Fe2+. Suprisingly, it was lately found that in the absence of TF, solute carrier family 39 member 14 (SLC39A14) directly mediates the passage of extracellular non transferrin bound iron across the cell membrane into the intracellular compartment and causes ferroptosis.

Due to the instability and high reactivity of Fe2+, excess Fe2+ generates hydroxyl radicals through Fenton reaction with hydrogen peroxide (H2O2), which directly reacts with polyunsaturated fatty acids (PUFAs) in cell membranes and plasma membranes to produce massive lipid ROS, Finally leading to cell death . Excess iron ions are stored through the formation of ferritin polymers , and Fe2+ is exported extracellularly through membrane ferroportin (FPN) , thus keeping iron level inside the cell in homeostasis. Ferritin is formed of 24 subunits of ferritin heavy chain 1 (FTH1) and ferritin light chain (FTL), which chelate approximately 4500 iron atoms. It was indicated that increasing ferritin break down or supressing ferritin expression increases intracellular LIP and increases cellular sensitivity to ferroptosis. In contrast, ferritin and its derivatives, and iron chelators helps ferroptosis resistance by decreasing intracellular iron ion levels or inhibiting the activity of several iron-containing metalloenzymes that catalyze lipid peroxidation reactions. SLC40A1-encoded FPN is the only known iron-exporting protein in mammals and is included in the Fe2+ efflux mechanism to maintain iron homeostasis and regulate ferroptosis. Ubiquitin-specific protease 35 (USP35) was discovered to interact directly with FPN and function as a deubiquitinating enzyme to maintain its protein stability. Whereas, USP35 knockdown elevates intracellular LIP levels and induces ferroptosis by reducing FPN-mediated iron export.

Ferroptosis in Autoimmune Hepatitis:

Microarray analysis indicated that ferroptosis may occur in mice with autoimmune hepatitis (AIH). S100-induced autoimmune hepatitis in a mouse model revealed that the knockdown of GPX4 increased the S100-induced accumulation of the lipid peroxide MDA and Fe2+ in liver tissues, hence significantly exacerbating ferroptosis in AIH. Fer-1 is a well-known and commonly used inhibitor of ferroptosis that has been shown to counteract S100-induced autoimmune hepatitis (AIH) and the resulting ferroptosis, thereby diminishing liver damage. This research aims to discover the importance of ferroptosis in immune-mediated hepatitis, suggests its potential role in the progression of autoimmune hepatitis as either an initiator or a mediator, and highlights the promise of targeting ferroptosis to enhance treatment options for JAIH, offering new insights for managing the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between one day and 18 years (children)
* patients diagnosed clinically and physically with juvenile autoimmune hepatitis including seronegative autoimmune hepatitis cases

Exclusion Criteria:

1. Cases with inadequate tissue in the paraffin block
2. Children with viral hepatitis
3. patients above the age of 18 years old

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases with adequate tissue in the paraffin blocks from Laboratories of Surgical Pathology at Assiut University and private labs will be recruited in this study during 5 years period from 2019 to 2024.
  Approximately 50 cases of juvenile autoimmune hepatitis and 10 control cases will be taken Histological diagnosis of H&E stained slides will be reviewed and the histological criteria will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Expression of USP35 in cases of juvenile autoimmune hepatitis | baseline
  Expression of USP35 is an indicator of ferroptosis so the investigators can detect the relationship between ferroptosis and the pathogenesis of juvenile autoimmune hepatitis

SECONDARY OUTCOMES:
To correlate the expression of USP35 with the level of necro-inflammation and extent of fibrosis using Massion's trichrome stain in cases of juvenile autoimmune hepatitis | baseline
  To know whether ferroptosis is an initiator or mediator in the pathogenesis of juvenile autoimmune hepatitis, the investigators will use Massion's trichrome stain to assess the level of neuroinflammation and extent of fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Howadya Ismail Hassan El Sayed, PhD, Study Director — Assiut University; Moemen Mostafa Ahmed Hafez, PhD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided